CLINICAL TRIAL: NCT00003398
Title: Evaluation of Allogeneic Marrow Transplants Depleted of T-Cells by CD34+ Selection in Patients Undergoing Transplantation With an Unrelated Matched or 1 Antigen Mismatched Donor or a 1 Antigen Mismatched Related Donor
Brief Title: Bone Marrow Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: UM Greenebaum Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000066400; MSGCC-9739; NCI-V98-1433
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Anemia; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; Burkitt lymphoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute eosinophilic leukemia; adult acute basophilic leukemia; adult acute megakaryoblastic leukemia (M7); childhood acute myeloblastic leukemia with maturation (M2); childhood acute promyelocytic leukemia (M3); childhood acute myelomonocytic leukemia (M4); childhood acute eosinophilic leukemia; childhood acute basophilic leukemia; childhood acute megakaryocytic leukemia (M7); stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; anemia; graft versus host disease; adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Anemia; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Basophilic, Acute; Leukemia, Megakaryoblastic, Acute; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Antilymphocyte Serum; Filgrastim; Cyclophosphamide; Thiotepa; Radiotherapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Drug: cyclophosphamide
Drug: thiotepa
Procedure: allogeneic bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Radiation: radiation therapy

SUMMARY:
RATIONALE: Bone marrow that has been treated to remove certain white blood cells may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy, and may reduce the chance of developing graft-versus-host disease following bone marrow transplantation.

PURPOSE: Phase IV trial to study the incidence of graft-versus-host disease in patients who have hematologic cancer and who are undergoing bone marrow transplantation from a donor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the incidence of acute graft versus host disease in patients undergoing transplantation with an unrelated or related matched or mismatched antigen donor. II. Evaluate the rapidity of engraftment and CD4 count recovery post-transplantation in this patient population.

OUTLINE: Patients receive total body irradiation (TBI) three or two times a day on days -8 to -5. Following TBI, patients receive thiotepa IV over 4 hours daily on days -4 and -3 plus cyclophosphamide IV over 1 hour daily on days -2 and -1. Antithymocyte globulin is administered by IV over at least 4 hours on days -4 to -1. Patients undergo an allogenic bone marrow transplantation on day 0. Bone marrow is harvested from patient's donor, depleted of T-cells, and infused. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 4.

PROJECTED ACCRUAL: Approximately 26-45 patients will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignancy or condition of the following types: Acute myelogenous leukemia (not M5 or M6) or lymphocytic leukemia in first or greater remission or early relapse OR Chronic myelogenous leukemia OR Myelodysplastic syndrome OR Aggressive or refractory non-Hodgkin's lymphoma OR Aggressive or refractory Hodgkin's disease OR Multiple myeloma at early relapse or after conventional chemotherapy to reduce tumor mass OR High risk chronic lymphocytic leukemia OR Aplastic anemia HLA-matched or 1 antigen mismatched (related or unrelated) available as donor

PATIENT CHARACTERISTICS: Age: 50 and under Performance status: Karnofsky 70-100% Life expectancy: Greater than 8 weeks Hematopoietic: Not specified Hepatic: Bilirubin less than 2 mg/dL SGOT less than 4 times upper limit of normal (ULN) Renal: Creatinine less than 2 times ULN OR Creatinine clearance greater than 60 mL/min Cardiovascular: LVEF at least 50% by MUGA Pulmonary: DLCO at least 50% Other: HIV negative No active extramedullary disease Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 1998-09; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry R. Meisenberg, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland, United States